CLINICAL TRIAL: NCT06636617
Title: Safety, Dosimetry and Treatment Response of 177Lu-JH04 in Patients with FAP-Positive Tumors
Brief Title: 177Lu-JH04 in Patients with FAP-Positive Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: FirstAHFujian-177Lu-JH04
Record Dates: First submitted 2024-09-22; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Patients with Advanced Metastatic FAP-Positive Tumors
Keywords: Lu-177; FAP; Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 3.70 GBq (100 mCi) of 177Lu-JH04 (Experimental): All 3 patients were intravenous injected with single dose 3.70 GBq (100 mCi) of 177Lu-JH04.
  Interventions: Drug: 3.70 GBq (100 mCi) of 177Lu-JH04
- 5.55 GBq (150 mCi) of 177Lu-JH04 (Experimental): All 3 patients were intravenous injected with single dose 5.55 GBq (150 mCi) of 177Lu-JH04.
  Interventions: Drug: 5.55 GBq (150 mCi) of 177Lu-JH04
- 7.40 GBq (200 mCi) of 177Lu-JH04 (Experimental): All 3 patients were intravenous injected with single dose 7.40 GBq (200 mCi) of 177Lu-JH04.
  Interventions: Drug: 7.40 GBq (200 mCi) of 177Lu-JH04

INTERVENTIONS:
Drug: 3.70 GBq (100 mCi) of 177Lu-JH04 — All 3 patients were intravenous injected with single dose 3.70 GBq (100 mCi) of 177Lu-JH04.
  Arms: 3.70 GBq (100 mCi) of 177Lu-JH04
Drug: 5.55 GBq (150 mCi) of 177Lu-JH04 — All 3 patients were intravenous injected with single 5.55 GBq (150 mCi) of 177Lu-JH04
  Arms: 5.55 GBq (150 mCi) of 177Lu-JH04
Drug: 7.40 GBq (200 mCi) of 177Lu-JH04 — All 3 patients were intravenous injected with single 7.40 GBq (200 mCi) of 177Lu-JH04
  Arms: 7.40 GBq (200 mCi) of 177Lu-JH04

SUMMARY:
This is a pilot study to assess the dosimetry, toxicity and response of 177Lu-JH04, a new FAP-targeted radiopharmaceutical, in patients with FAP-Positive Tumors. All patients underwent 68Ga-FAPI PET/CT for selection and were successively divided into three groups of 3 people each.The three groups received successively an approximately 3.70 GBq (100 mCi), 5.55 GBq (150 mCi) and 7.40 GBq (200 mCi) of 177Lu-JH04 up to 4 cycles.

DETAILED DESCRIPTION:
Cancer-associated fibroblasts (CAFs) are an integral part of the tumor microenvironment and present abundantly in the stroma of multiple tumor entities. Fibroblast activation protein (FAP), as a specific marker protein of CAFs, is overexpressed on more than 90% of malignant tumors& limited and expression in normal tissues, making it an appropriate target for diagnosis and therapy of numerous malignant tumors. Currently, several radiopharmaceuticals targeting FAP for radionuclide therapy have been developed, such as 177Lu-FAPI-46, 177Lu-FAP-2286, and showed high efficacy and reasonable toxicity profile in tumor treatment. 177Lu-JH04, a novel radiopharmaceutical targeting FAP, demostrated high stability in vitro and in vivo, and can accumulate specifically in tumors with high binding affinity, safety, and selectivity in preclinical studies. In this study, we assess the dosimetry, toxicity and response of 177Lu-JH04 for the treatment of patients with advanced metastatic cancers after exhaustion of all other treatment options.

ELIGIBILITY:
Inclusion Criteria:

* progressive advanced metastatic tumors
* tumors with high FAP expression confirmed on 68Ga-FAPI PET/CT
* adequate renal, haematological, and liver function
* an Eastern Cooperative Oncology Group performance status of 0-2

Exclusion Criteria:

* pregnant or lactating women
* received other radionuclide therapy in the past 6 months
* received chemotherapy, radiotherapy and other anti-tumor treatments in the past 28 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Toxic and side effect | through study completion, an average of 2 weeks
  The white blood cell count, granulocyte count, platelet count, hemoglobin count and serum biochemicals of each patient before and after each treatment were recorded and compared. And the weight (in kilograms) of the patients was monitored. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Dosimetry of normal organs and tumors | through study completion, an average of 4 weeks
  The semiquantitative dosimetry will be performed based on SPECT/CT acquisitions after the first administration of 177Lu-JH04. The dose delivered to normal organs and tumors will be recorded.

OTHER OUTCOMES:
Treatment Response | through study completion, an average of 3 months
  The number and size (long diameter in centimeter) of tumors were calculated and compared based on enhanced CT and MRI. The treatment effect of tumors was evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — The First Affiliated Hospital, Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China